CLINICAL TRIAL: NCT07138157
Title: Comparison Of The Effects Of Two Different Exercise Training Based On Internal And External Focus In Children and Adolescents With Rheumatic Diseases
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Aleyna Yilmaz, Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbuIUC
Record Dates: First submitted 2025-06-29; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Juvenile Dermatomyositis; Rheumatic Diseases; Juvenile Idiopathic Arthritis (JIA); Familial Mediterranean Fever (FMF)
Keywords: Juvenile dermatomyositis; Exercise in pediatric rheumatic diseases; External focus; Internal focus
MeSH Terms: conditions — Dermatomyositis; Rheumatic Diseases; Arthritis, Juvenile; Familial Mediterranean Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Focus of Attention Group (Active Comparator): In this group, the exercise program will be implemented using external focus in the commands and exercise instructions. During exercise, external focus commands are designed to direct attention toward the impact of the movement or an external stimulus. For example, during the squat exercise, the command "Bend over as if sitting on a chair until the sign in front is no longer visible" represents an external focus command, whereas the command "Bend over by bending the knees without disturbing the straightness of the back" represents an internal focus command.
  Interventions: Other: External Focus Exercises
- Internal Focus of Attention Group (Active Comparator): In this group, the exercise program will be implemented using internal focus in the commands and exercise instructions. During exercise, internal focus commands are designed to direct attention toward the body part performing the movement or the movement itself. For example, during the squat exercise, the command "Bend over by bending the knees without disturbing the straightness of the back" represents an internal focus command, whereas the command "Bend over as if sitting on a chair until the sign in front is no longer visible" represents an external focus command.
  Interventions: Other: Internal Focus Exercises

INTERVENTIONS:
Other: External Focus Exercises — The commands given during the exercises will encourage the participants to focus their attention on the effect of the movement/ external focus of attention
  Arms: External Focus of Attention Group
Other: Internal Focus Exercises — The commands given in the second group will encourage the participants to focus their attention on the body part performing the movement/ Internal focus of attention
  Arms: Internal Focus of Attention Group

SUMMARY:
The study aims to compare the effects of two different exercise programs, based on distinct focus strategies, on physical fitness and fatigue in children and adolescents with rheumatic diseases. Participants will include individuals diagnosed with Juvenile Idiopathic Arthritis (JIA), Juvenile Dermatomyositis (JDM), and Familial Mediterranean Fever (FMF), monitored at Istanbul University, Istanbul Faculty of Medicine, in collaboration with Istanbul University-Cerrahpaşa, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation. After baseline assessments, participants will be randomly allocated into two groups. One group will receive an exercise program with commands and instructions emphasizing external focus, while the other group will follow a program emphasizing internal focus. Both exercise interventions will last for 8 weeks, consisting of two online supervised sessions and one home-based session per week under family supervision. Final evaluations will be conducted at the clinic after completion of the intervention period.

DETAILED DESCRIPTION:
Juvenile Idiopathic Arthritis (JIA), Juvenile Dermatomyositis (JDM) and Familial Mediterranean Fever (FMF) patients who were monitored at Istanbul University Istanbul Faculty of Medicine under the supervision of Istanbul University-Cerrahpaşa, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation will be included in this study. Demographic data of the participants, including age, weight, height, body mass index, age of onset of the disease, time elapsed before diagnosis, duration of symptoms, family history, will be recorded. Participants' physical fitness, muscle strength and functions, physical activity levels, fatigue and pain levels will be evaluated face-to-face at the beginning and at the end of the 8-week exercise program. The FitnessGram test battery will be used for the physical fitness assessment. The 'Fatigue Severity Scale' will be used to assess the fatigue levels of the participants. Physical activity levels will be evaluated separately in children and adolescents using the 'Physical Activity in Adolescents Questionnaire' and the 'Physical Activity in Children Questionnaire'. In all cases, pain severity will be questioned using the 'Visual Analog Scale'. All participants will be given a 6 Minute Walk Test to measure their functional capacity, 30 Seconds Sit to Stand Test to measure their lower extremity strength.

Following to first evaluation, the patients will be randomly assigned to two groups. In the first group, the exercise program will be applied as the basis of external focus in the commands and exercise instructions directed to the patient, while in the second group, the exercise program will be applied as the basis of internal focus. Exercise training in both groups lasted 8 weeks; It will be applied 3 days a week, two sessions each week under the supervision of an online physiotherapist and one session with online family supervision. Online training sessions will be conducted via Google Meets. In the first group, the exercise program will be applied based on the external focus, while in the second group, the exercise program will be applied on the basis of the internal focus. The same exercise program will be applied in both groups, but in the first group, the commands given during the exercises will encourage the participants to focus their attention on the effect of the movement, while the commands given in the second group will encourage the participants to focus their attention on the body part performing the movement. In the squat exercise, for instance, the first group is instructed to "Bend over as if sitting on a chair until the sign in front is no longer visible" represents an external focus command, whereas the command "Bend over by bending the knees without disturbing the straightness of the back" represents an internal focus command.

Exercise training in both groups last 8 weeks; two sessions each week online via Google Meets and third session will be held under family supervision. At the end of 8 weeks, participants will be called back to the clinic for a final evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile Dermatomyositis: Being diagnosed with JDM according to the Bohan and Peter Criteria by a pediatric rheumatologist
* Familial Mediterranean Fever: Having been diagnosed with FMF at least 6 months ago
* JIA: Having been diagnosed with JIA according to the ILAR classification
* Not having visual impairment or hearing impairment
* Being at a mental level that can adapt to the exercise program
* Having internet connection

Exclusion Criteria:

* Having any systemic chronic disease other than JIA, FMF, or JDM
* Having any musculoskeletal disease or an orthopedic, neurological, psychological disease that may interfere with participation in exercise
* Having developed amyloidosis
* Having undergone surgery affecting the musculoskeletal system in the last 6 months
* Having visual impairment or hearing impairment
* Not having internet connection

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Fitness | 8 weeks
  Overall physical fitness will be assessed using the FitnessGram Physical Activity Test Battery, a validated tool for evaluating health-related fitness components in children and adolescents. The battery includes subtests to measure cardiovascular endurance (PACER test), muscular strength and endurance (curl-up, push-up), and flexibility (sit-and-reach). Each subtest will be scored separately according to criterion-referenced health standards established for children and adolescents. Changes in performance scores from baseline to 8 weeks will be analyzed to determine the effectiveness of the intervention on physical fitness.
Change in Fatigue Severity | 8 weeks
  Fatigue severity will be assessed using Fatigue Severity Scale (FSS), which is validated tools for measuring perceived fatigue intensity and its impact on daily functioning. The FSS comprises nine items rated on a 7-point Likert scale, with a mean score ≥4 considered indicative of substantial fatigue. The change from baseline to post-intervention will be analyzed. This outcome will provide a quantitative evaluation of the intervention's effectiveness in mitigating clinically relevant fatigue in the target population.
Change in Pain Intensity | 8 weeks
  Pain intensity will be evaluated using the Visual Analog Scale (VAS), a reliable and validated tool commonly used in both clinical and research settings. Participants will be asked to rate their pain on a 10 cm horizontal line, where 0 cm indicates "no pain" and 10 cm represents "worst imaginable pain." A decrease of at least 2 cm is generally considered to be clinically meaningful. Changes in VAS pain scores from baseline to the end of the intervention will be analyzed to determine the intervention's impact on pain.

SECONDARY OUTCOMES:
Change in Physical Activity Level (Children) | 8 weeks
  Physical activity level will be assessed using the Physical Activity Questionnaire for Children (PAQ-C) for participants aged 8-14 years. This questionnaire is self-administered, 7-day recall instruments that generate a composite score ranging from 1.00 to 5.00, where higher scores indicate higher levels of physical activity. Scores between 1.00 and 2.33 are generally interpreted as low activity, 2.34 to 3.66 as moderate activity, and 3.67 to 5.00 as high activity. The change in PAQ-C scores from baseline to post-intervention will be analyzed.
Change in Physical Activity Level (Adolescents) | 8 weeks
  Physical activity level will be assessed using the Physical Activity Questionnaire for Adolescents (PAQ-A) for participants aged 14-18 years. This is a self-administered, 7-day recall instrument that generates a composite score ranging from 1.00 to 5.00, with higher scores indicating higher levels of physical activity. Scores between 1.00 and 2.33 are interpreted as low activity, 2.34 to 3.66 as moderate activity, and 3.67 to 5.00 as high activity. Changes in PAQ-A scores from baseline to 8 weeks will be analyzed.
Change in Functional Capacity | 8 weeks
  Functional capacity will be assessed using the 6-Minute Walk Test (6MWT), a widely used and validated measure of submaximal exercise performance in pediatric populations. The test evaluates the total distance walked on a flat surface within six minutes, reflecting the individual's ability to perform daily physical activities. Changes in walking distance from baseline to 8 weeks will be analyzed to determine the effectiveness of the exercise program on functional capacity.
Change in Lower Extremity Strength | 8 weeks
  Lower extremity strength will be assessed using the 30-Second Sit-to-Stand Test. The test evaluates the number of sit to stand repetitions in 30 seconds reflecting the individual's lower extremity strength. Changes in repetitions from baseline to 8 weeks will be analyzed to determine the effectiveness of the exercise program on lower extremity strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No